CLINICAL TRIAL: NCT05048940
Title: Randomized, Open-label, Adaptive, Controlled, Phase III Clinical Trial to Evaluate the Efficacy, Safety and Immunogenicity of Reimmunization With Third Dose of Homologous vs. Heterologous Vaccine Against COVID-19 in Patients Undergoing Solid Organ Transplantation: Liver, Heart, Kidney and Lung.
Brief Title: Efficacy, Safety, and Immunogenicity of Vaccine Reimmunization With a Third Homologous Versus Heterologous Dose Against COVID-19 in Patients Undergoing Solid Organ Transplantation.
Acronym: REIN-TX
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The health authority indicates that the official vaccination schedule differs from that described in the protocol.
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REIN-TX
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Covid19
Keywords: Vaccine; Covid-19; Liver Trasplant; Lung Trasplant; Heart Trasplant; Kidney Trasplant
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HETEROLOGOUS VACCINE (Experimental): COVID-19 Vaccine Janssen, injectable suspension
  Interventions: Biological: Janssen vaccine
- HOMOLOGOUS VACCINE (Active Comparator): Spikevax (Moderna), injectable dispersion
  Interventions: Biological: Spikevax (Moderna) vaccine

INTERVENTIONS:
Biological: Janssen vaccine — 0.5 ml millilitre(s) Intramuscular use
  Other Names: Janssen Biologics B.V.; EU/1/20/1525/001 EU/1/20/1525/002
  Arms: HETEROLOGOUS VACCINE
Biological: Spikevax (Moderna) vaccine — 0.5 ml millilitre(s) Intramuscular use
  Other Names: MODERNA BIOTECH SPAIN, S.L.; EU/1/20/1507/001
  Arms: HOMOLOGOUS VACCINE

SUMMARY:
Patients undergoing solid organ transplantation randomly selected from those who have received two doses of Spikevax (Moderna) vaccine, provided that a minimum of 8 weeks have elapsed from the second dose to the time of the start of the trial. It is planned to include 386 patients.

DETAILED DESCRIPTION:
The main objective of this trial is to evaluate the immunogenicity of reimmunization against SARS-CoV-2 in patients undergoing solid organ transplantation with heterologous revaccination, testing whether in patients who received two doses of Spikevax Moderna vaccine there is a significant increase at 28 days in their antibody titers against SARS-CoV-2 after receiving a dose of Janssen.

The secondary objectives of this trial are:

1. To evaluate the efficacy of reimmunization against SARS-CoV-2 in subjects undergoing solid organ transplantation, in terms of incidence of infection and severity of COVID-19 after revaccination in the transplanted patient.
2. To gain insight into the humoral and cellular immune response conferred by the sequential combination of both homologous and heterologous vaccination over one year, as well as its duration in subjects undergoing solid organ transplantation.
3. To evaluate the safety of vaccines against SARS-CoV-2 in subjects undergoing solid organ transplantation.
4. To determine the potential existence of differences in humoral (Anti S Ac) and cellular immune response depending on the immunosuppression regimen.
5. To evaluate the occurrence of side effects, including rejection and anti-HLA and DSA antibodies after revaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent solid organ transplantation prior to revaccination against COVID-19.
2. Patients who have received the full COVID-19 vaccination regimen with Spikevax (Moderna) vaccine, with a minimum of 8 weeks having elapsed from the second dose to the time of trial initiation.
3. Age > 18 years.
4. All participants must have previously agreed to participate in the study by signing the informed consent form.

Exclusion Criteria:

1. Having suffered SARS-CoV-2 infection at any time prior to inclusion in the study.
2. Subjects without solid organ transplantation or with a different solid organ (e.g. pancreas transplantation) and without any type of immunosuppression (immunocompetent non-transplanted) from the general population.
3. Age < 18 years
4. Temperature of at least 38°C in the 24 hours prior to immunization or other clinically relevant acute symptomatology.
5. Clinical manifestations compatible with COVID-19 infection at the time of evaccination.
6. Known allergy or history of anaphylaxis or other serious adverse events to the administration of vaccines or their excipients.
7. Any other condition that contraindicates vaccination against SARSCov2, including pregnancy.
8. Having presented graft rejection in the 15 days prior to the start of the study.
9. Any condition or situation that may interfere with the ability to maintain adherence to study procedures and visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the production of anti-S1-RBD IgG antibodies. | 28 days
  Positivity for comparison before and after revaccination and according to homologous or heterologous vaccination will be quantified in the laboratory method units.

SECONDARY OUTCOMES:
Change in the presence of activated T cells specific for SARS-CoV-2 (Sprotein). | 1 year
  T-cell response to SARS-CoV-2 will be analyzed by flow cytometry.
Changes in the phenotype of effector/memory/virgin B and T cell populations and subtypes of Th and NK cell populations. | 1 year
  T-cell response to SARS-CoV-2 will be analyzed by flow cytometry.
Incidence of symptomatic/asymptomatic COVID infection after revaccination. | 1 year
  Confirmed COVID-19 is defined as the presence of at least one of the following symptoms: fever, new onset or increased cough, new onset or increased shortness of breath, chills, new onset or increased muscle pain, loss of taste or smell, sore throat, diarrhea or vomiting, combined with a respiratory specimen, obtained during the symptomatic period, positive for SARS-CoV-2 by nucleic acid amplification (PCR)-based testing or antigen testing.
Number of patients with hospital admissions and/or visits to the emergency department for severe symptoms related to COVID-19 infection. | 1 year
  Confirmed COVID-19 is defined as the presence of at least one of the following symptoms: fever, new onset or increased cough, new onset or increased shortness of breath, chills, new onset or increased muscle pain, loss of taste or smell, sore throat, diarrhea or vomiting, combined with a respiratory specimen, obtained during the symptomatic period, positive for SARS-CoV-2 by nucleic acid amplification (PCR)-based testing or antigen testing.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Crespo García, Principal Investigator — Hospital Universitario Marqués de Valdecilla; Marcos López Hoyos, Principal Investigator — Hospital Universitario Marqués de Valdecilla
Locations (1):
- Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain